CLINICAL TRIAL: NCT00878839
Title: Investigation of Corneal Aberrations and Visual Outcomes in Patients Implanted With an AcrySof Toric Intraocular Lens (IOL)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Product availability
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M09-016
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-06

CONDITIONS: Cataracts; Astigmatism
Keywords: Cataract; Toric IOL; Corneal Aberration; Astigmatism; AcrySof
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Toric (Other): AcrySof Toric IOL to assess corneal aberration
  Interventions: Device: Toric

INTERVENTIONS:
Device: Toric — AcrySof Toric IOL

SUMMARY:
A prospective evaluation of postoperative corneal aberrations and visual parameters (e.g. visual acuity) in patients implanted with an AcrySof Toric IOL.

ELIGIBILITY:
Inclusion Criteria:

* Operable cataracts;
* Good ocular health;
* Qualifies for AcrySof Toric IOL via AcrySof Toric Calculator (1.03-2.06 D cylinder at corneal plane)

Exclusion Criteria:

* >2.06 D astigmatism at corneal plane;
* irregular astigmatism;
* prior or ongoing corneal disease or scarring;
* history of ocular disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Corneal Aberration | 3 months

SECONDARY OUTCOMES:
Visual acuity, residual refractive cylinder, lens alignment | 3 months